CLINICAL TRIAL: NCT03980860
Title: Effect of HIIT vs Low Intensity Training on Fat Loss in Obese Patients
Brief Title: Effect of Two Exercise Programs on Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Adarsh Gupta, DO, MS, FACOFP, Professor of Family Medicine, Rowan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2019000482
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: This is a case/control study comparing overweight/obese patients of three different groups (control, HIIT, LIT). The goal of a case/control is to show whether exposure to HIIT, two times a week for 6 weeks will decrease lean body mass versus control and LIT. If it turns out that lean body mass does decrease, then HIIT is not an effective exercise modality for overweight/obese patients, and in fact LIT or control may be a better option.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT (High Intensity Interval Training) (Active Comparator): Subjects are undergoing high intensity interval training
  Interventions: Other: Exercise Type
- Low intensity training long duration (Active Comparator): Subjects are undergoing a lower intensity training program for a long duration
  Interventions: Other: Exercise Type
- Control (No Intervention): No exercise program intervention (usual care)

INTERVENTIONS:
Other: Exercise Type — The implementation of 2 types of exercise programs to reduce body fat
  Arms: HIIT (High Intensity Interval Training); Low intensity training long duration

SUMMARY:
The purpose of the study is to compare the effectiveness of two exercise programs (High Intensity Interval Training/HIIT and Low Intensity (LIT) Long Duration training) on decreasing fat mass and preserving lean body mass in obese patients. What the investigators are proposing is that HIIT is less effective because it will most likely decrease lean body mass in obese patients, whereas LIT decreases fat mass and conserves lean body tissue.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with a BMI of 25 and above

Exclusion Criteria:

* Those that cannot exercise

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Body fat | 6 weeks
  Reduction in body fat
Lean body mass | 6 weeks
  Retention of lean body mass

SECONDARY OUTCOMES:
Blood pressure | 6 weeks
  Reduction of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh Gupta, DO, Principal Investigator — Rowan University
Locations (1):
- Rowan SOM Family Medicine, Stratford, New Jersey, United States